CLINICAL TRIAL: NCT07103174
Title: A Phase II Clinical Study on the Efficacy and Safety of MG-K10 Humanized Monoclonal Antibody Injection in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of MG-K10 Humanized Monoclonal Antibody Injection in Subjects With Atopic Dermatitis
Acronym: MG-K10
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Mabgeek Biotech.Co.Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MG-K10-AD-005
Record Dates: First submitted 2025-06-30; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MG-K10 Regimen 1 (Experimental): Administer the drug once every 4 weeks for a total of 6 times
  Interventions: Biological: MG-K10 placebo
- MG-K10 Regimen 2 (Active Comparator): Administer the drug once every 4 weeks for a total of 6 times
  Interventions: Biological: MG-K10 placebo

INTERVENTIONS:
Biological: MG-K10 placebo — Administer the drug once every 4 weeks for a total of 6 times

SUMMARY:
This study is a multicenter, randomized, double-blind, parallel controlled phase II study. It is planned to include approximately 60 subjects with moderate to severe atopic dermatitis(AD) to evaluate the efficacy and safety of MG-K10 monotherapy in adult patients with moderate to severe AD, and to observe PK characteristics, PD effects and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. AD patients diagnosed in accordance with the consensus criteria of the American Academy of Dermatology (2014) had a history of AD or eczema diagnosis of ≥1 year
2. The patient's response to topical medication treatment is insufficient, or it is medically inappropriate to use topical medication for treatment
3. The subjects and their partners agreed to take effective contraceptive measures from signing the Informed Consent Form (ICF) until 6 months after the end of treatment, and had no plans for childbirth, sperm donation or egg donation

Exclusion Criteria:

1. The subject currently has a diagnosis of other active skin diseases (such as psoriasis or lupus erythematosus) that may affect the evaluation of AD
2. Patients with eye diseases that the researchers judged as unsuitable for inclusion
3. Patients with malignant tumors within 5 years
4. There is evidence of active tuberculosis, or there has been evidence of active tuberculosis before and no appropriate documented treatment has been received
5. Confirm active parasitic infection
6. Those with active hepatitis, or positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb), or positive for hepatitis C virus (HCV) antibody, or positive for HIV antibody, or positive for (TP-Ab)
7. Women who are breastfeeding or pregnant, or women planning to become pregnant or breastfeed during the study period
8. Those who the researchers consider to have other circumstances that make them unsuitable to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-16 (Estimated); Primary Completion 2027-07-16 (Estimated); Study Completion 2027-12-16 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects reaching EASI-75 at 24 weeks of treatment | 24 weeks
  The percentage of subjects reaching EASI-75 at 24 weeks of treatment
The percentage of subjects who achieved the IGA score standard at 24 weeks of treatment | 24 weeks
  The percentage of subjects whose IGA score reached 0 or 1 at 24 weeks of treatment (W24) and decreased by ≥2 points compared with the baseline;

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tower 5,No.34,Chunxiao Road No.122 Pudong District, Shanghai, 201203.p R. china, Shanghai, Shanghai Municipality
  - Hangzhou First People's Hospital, Zhejiang, 杭州

IPD SHARING:
Plan to Share IPD: No